CLINICAL TRIAL: NCT06059495
Title: Watch-and-wait Strategy to Initiate Dostarlimab-based Immunotherapy in Localized Deficient Mismatch Repair (dMMR) and/or Microsatellite Instability High (MSI-H) oEso-gastric Junction and Gastric Adenocarcinoma: An Open-label GERCOR Phase II Study
Brief Title: Watch-and-Wait Approach With Dostarlimab in Localized dMMR/MSI-H Gastric Cancer: GERCOR Phase II Study
Acronym: DEWI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEWI G-123; 2023-506102-39-00 (Other: EU CT)
Record Dates: First submitted 2023-07-20; First posted 2023-09-28 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Adenocarcinoma - GEJ; Gastric Adenocarcinoma
Keywords: dMMR; MSI-H; dostarlimab; watch-and-wait; surgery; immunotherapy
MeSH Terms: interventions — dostarlimab

STUDY DESIGN:
Intervention Model Description: After inclusion all patients will receive dostarlimab at 500 mg q3w (± 2-3 days) for 4 cycles (C1-C4).
  An adaptive treatment strategy will be determined based on clinical assessment of the patient at weeks 12 (±1 week) and week 24 (±1 week).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dostarlimab-based treatment (Experimental): After inclusion patients will receive dostarlimab at 500 mg q3w (± 2-3 days) for 4 cycles (C1-C4). Then, an adaptive treatment strategy will be determined based on clinical assessment of the patient.
  Interventions: Drug: Dostarlimab

INTERVENTIONS:
Drug: Dostarlimab — After inclusion: dostarlimab 500mg IV 30min q3w (± 2-3 days) for 4 cycles (C1-C4)
  Then:
  At wk12 • If cCR: dostarlimab 1000mg q6w for 2 cycles (C5-C6)
  • If downstaging at UGI endoscopy, and no disease progression (PD)/or mets on TAP-CT, <3 biopsies with tumor cells: dostarlimab 500mg q3w for 4 cycles (C5-C8)
  • If loco/loco-regional PD on TAP-CT, macroscopic tumor on UGI endoscopy, no distant mets, and >2 positive biopsies at wk12 followed by surgery and if Becker-TRG 1a, 1b, or 2 after surgery: dostarlimab 1000mg q6w for 6 cycles (C5-C10)
  At 24wk
  • If cCR at 12 and 24 wks: dostarlimab 1000mg q6w for 4 cycles (C7-C10)
  • If downstaging at UGI endoscopy without PD on CT at wk 12 with <3 biopsies with tumor cells at wk12 and cCR: dostarlimab 1000mg q6w for 4 cycles (C9-C12)
  • If downstaging at UGI endoscopy without PD on CT at wk 12 with and no cCR, surgery will be proposed and if Becker-TRG 1a, 1b, or 2 after surgery: dostarlimab 1000mg q6w for 4 cycles (C9-C12)
  Other Names: Jemperli

SUMMARY:
This phase II study will evaluate dostarlimab with a watch-and-wait approach for patients with localized mismatch repair deficiency (dMMR)/microsatellite instability (MSI) gastric or oeso-gastric junction adenocarcinoma.

The goal of the study is to determine whether the surgery could be avoided in patients with localized dMMR/MSI-H gastric/OGJ adenocarcinoma with complete response at endoscopy and biopsies free of tumoral cells after treatment with dostarlimab, with a watch-and-wait approaches.

DETAILED DESCRIPTION:
In patients with localized, resectable gastric or oeso-gastric junction (OGJ) adenocarcinoma radical surgery is the only curative option. Despite the evolution in treatment with multimodality strategies, gastric or OGJ adenocarcinoma remains one of the most lethal malignancies. When the disease is localized, perioperative chemotherapy with cytotoxic agents is the preferred strategy.

The morbidity rate associated with oesophagogastrectomy/gastrectomy and their negative impact on patients' quality of life and considering the high efficacy of ICIs in patients with localized tumor, one might wonder whether the surgery could be avoided in patients with localized dMMR/MSI-H gastric/OGJ adenocarcinoma

The purpose of this national, multicenter, open-label phase II study is to look at the effects of the immunotherapy drug dostarlimab with a watch-and-wait approach in patients with localized dMMR/MSI gastric or oeso-gastric junction adenocarcinoma and to determine whether patients with complete response at endoscopy and biopsies free of tumoral cells after treatment with dostarlimab, with a watch-and-wait approach can circumvent surgical resection.

The primary objective of the study is the rate of complete clinical response at 1 year.

A total of 59 patients are expected to be enrolled in the study. Patients will be included in participating centers, which will perform treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed and dated informed consent,
2. An ECOG PS of 0-1,
3. ≥18 and ≤75 years old,

   The patient over 75 years of age is eligible only if all the following conditions are met:
   * The patient's G8 questionnaire score is above 14 AND
   * The patient is eligible for surgery and has no contraindications to repeated UGI endoscopy with biopsies,
4. Histologically proven non-metastatic gastric or OGJ adenocarcinoma cT2 to T4, Nx, M0 after computed tomography thorax-abdomen-pelvis (TAP-CT) and echo-endoscopy (EUS) according to the 7th Edition of the International Union Against Cancer; NB: Echo-endoscopy will be performed only if the tumor is not obstructive at UGI endoscopy ± a new UGI endoscopy with 10 biopsies, photos (if not done at the first UGI endoscopy done for diagnosis) and if possible (not mandatory) tumor tattooing/inking. If obstructive, the tumor will be classified as cT3 or cT4 (in the situation when the tumor was obstructive and prevented EUS, it was classified T3N+, if it did not invade the adjacent organs on CT scan, because obstructing tumours represented locally advanced disease in the vast majority of cases in previous studies). In this case a new UGI endoscopy must be done with 10 biopsies, photos (if not done at the first GGI endoscopy done for diagnosis) and if possible (not mandatory) tumor tattooing/inking to follow the location of the tumor.
5. No peritoneal carcinomatosis (optional coelioscopy; recommended in case of doubt/ suspicious on CT/ imaging),
6. No prior therapy (chemotherapy, radiotherapy, or immunotherapy) for localized gastric or OGJ adenocarcinoma,
7. Tumor status confirmed to be dMMR/MSI-H as follows:

   - MMR protein expression status will be evaluated by immunohistochemistry (IHC) with four antibodies (anti-hMLH1, anti-hMSH2, anti-hMSH6, anti-hPMS2) according to the local procedures. dMMR will be defined as loss of MLSH1 and PMS2, loss of MSH2 and MSH6, or loss of only one protein with presence of MSI-H.

   MSI analysis will be performed by polymerase chain reaction [PCR] using a pentaplex panel (BAT-25, BAT-26, NR-21, NR-24, and NR-27; PROMEGA). MSI-H is defined as instability in two or more of the five studied markers. For the purpose of this study samples with 2 unstable markers will also undergo MMR analysis by IHC. Agreement of Sponsor (GERCOR) on a dMMR/MSI status is mandatory to include the patient (the patient's file [an anonymized mail] has to be send to Sponsor). Approval/refusal email for inclusion of the patient will be send by the Sponsor within 24 hours of receipt of the Investigator email. In case of discrepancy between IHC and PCR, the final decision about the dMMR/MSI status will be taken by GERCOR or coordinating investigator,
8. Hematological status: absolute neutrophil count (ANC) ≥1.5 x 109/L; platelets ≥100 x 109/L; hemoglobin ≥9 g/dL,
9. Adequate renal function: serum creatinine level ≤150 μM and clearance ≥50 ml/min (Modification of the Diet in Renal Disease [MDRD] or Cockcroft and Gault),
10. Adequate liver function: ≤1.5 x upper limit of normal (ULN) of direct bilirubin ≤ ULN for participants with total bilirubin levels >1.5 x ULN (inclusion possible if known Gilbert syndrome), alkaline phosphatase <5 x ULN, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤2.5 x ULN,
11. International normalized ratio (INR), prothrombin time (PT), and activated partial thromboplastin time (aPTT) ≤1.5 x ULN, except for the patient on anticoagulant therapy who must have PT-INR-aPTT within therapeutic range is deemed appropriate by the Investigator,
12. Radiological tumor assessment at screening performed within 28 days before inclusion according to RECIST version 1.1 by chest, abdomen, and pelvis CT, showing the absence of metastatic or non-surgical disease,
13. A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies:

    * Is a woman of non-childbearing potential as defined: i/ ≥ 45 years of age and has not had menses for >1 year, ii/ Amenorrheic for <2 years without a hysterectomy and oophorectomy and have a follicle stimulating hormone (FSH) value in the postmenopausal range upon pre-study (screening) evaluation, iii/ post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound, magnetic resonance imaging (MRI), or CT scan. Tubal ligation must be confirmed with medical records of the actual procedure, otherwise the patient must fulfill the criteria in Inclusion criteria 15. Information must be captured appropriately within the site's source documents,
    * Negative pregnancy blood test within 72 hours before the first dose of dostarlimab, AND
    * If woman of childbearing potential (WOCBP), female patient must be willing to use a highly effective form of contraception from screening throughout the study treatment and 4 months after the last dose of dostarlimab,
14. Male participants are eligible to participate if they agree to the following during the study treatment and for 4 months after the last dose of dostarlimab:

    * Refrain from donating sperm,
    * Must use contraception/barrier as follows:

      * Agree to use a male condom when having sexual intercourse with a WOCBP who is not currently pregnant.
      * Agree to use a male condom when engaging in any activity that allows for passage of ejaculate to another person,
15. Providing primary tumor tissue samples (processed as formalin-fixed, paraffin-embedded [FFPE] blocks or freshly frozen) acquired during UGI endoscopy together with images (mandatory), NB: The patient's agreement will be specifically requested for endoscopic images in the patient information note and informed consent for their use as clinical data that may be analyzed and presented in publications. These data will be used in the same manner as other personal data. The confidentiality of these data will be maintained,
16. Willingness and capablility to comply with scheduled visits, treatment schedule, laboratory tests, tumor biopsies, and other requirements of the study,
17. Registration in a National Health Care System (PUMa - Protection Universelle Maladie included).

Exclusion Criteria:

1. Prior concomitant unplanned antitumor therapy (e.g., chemotherapy, molecular targeted therapy, immunotherapy),
2. Treatment with any investigational medicinal product within 28 days prior to study entry,
3. Treatment anticoagulant or hemostasis disorder contraindicating - biopsies during endoscopy,
4. Major surgical procedure within 28 days (4 weeks) prior to the first dose of study treatment,
5. Other serious and uncontrolled non-malignant disease (including active infection) or is considered a poor medical risk due to a serious, uncontrolled medical disorder, nonmalignant systemic disease or active infection requiring systemic therapy. Specific examples include, but are not limited to, active, non-infectious pneumonitis; uncontrolled ventricular arrhythmia; recent (within 90 days) myocardial infarction; uncontrolled major seizure disorder; unstable spinal cord compression; superior vena cava syndrome; or any psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study,
6. Other concomitant or previous malignancy other than the disease under study, except as noted below:

   i/ adequately treated in-situ carcinoma of the uterine cervix, ii/ basal or squamous cell carcinoma of the skin, iii/ cancer from which the patients was in complete remission for ≥3 years,
7. Metastases (M stage disease) whatever the location,
8. Pregnancy or breastfeeding,
9. Human immunodeficiency virus (HIV),
10. Active hepatitis B virus (HBV, defined as having a positive hepatitis B surface antigen [HBsAg] test) or hepatitis C virus (HCV) prior to inclusion, Note: Patients with past HBV infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen antibody test) are eligible.

    Note: Patients positive for HCV antibody are eligible only if PCR testing is negative for HCV RNA.
11. Patient under a legal protection regime (guardianship, curatorship, judicial safeguard) or administrative decision or incapable of giving his/her consent,
12. Impossibility of submitting to the medical follow-up of the study for geographical, social, or psychiatric illness.

Non-eligible to immunotherapy:

1. Pyloric tumor, NB: tumors of the pylorus will be excluded because of the risk of high occlusion in case of pseudo progression and associated surgery,
2. Any history of autoimmune disease including, but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis, Note: History of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible.

   Note: Controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible.
3. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest imaging,
4. Any live, attenuated vaccine within 14 days prior to the firs dose of study treatment or such administration is anticipated during the study,
5. Prior therapy with any immune-checkpoint inhibitors, including antibodies or drugs targeting CD137, CTLA-4, PD-1, or PD-L1 or other checkpoint pathways,
6. Prior allogeneic bone marrow transplantation or prior solid organ transplantation,
7. Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within 2 weeks prior to the first dose of adjuvant treatment or is required to receive systemic immunosuppressive medications during the study. Inhaled or topical steroids and adrenal replacement doses >10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.

Note: Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled into the study after approval of the Medical Contact. Note: Subjects are permitted the use of topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Adrenal replacement steroid doses including doses >10 mg daily prednisone is permitted. A brief (less than 3 weeks) course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by a contact allergen) is permitted.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Clinical complete response (cCR) | From the start of therapy with dostarlimab to 1 year; assessed at 1 year.
  The primary endpoint is the rate of patients who at 1 year from the start of therapy with dostarlimab are alive, were not operated for tumor resection, are free of disease progression (locoregional or metastases), have all biopsies negative, and show endoscopy downstaging stage 3 and 4.

SECONDARY OUTCOMES:
Pathological complete response (pCR) | up to 5 years; from the date of dostarlimab initiation to the date of surgery
  Pathological complete response is defined as 100% fibrosis or fibro-inflammation or necrosis or granulomatous reaction within an entire gross lesion without microscopic evidence of carcinoma, and no positive lymph nodes, after examination of the complete macroscopic surgical specimen equivalent to a Becker TRG Grade 1a (complete regression).
Loco/loco-regional and distant recurrence | up to 5 years; from the date of dostarlimab initiation to the date of recurrence
  Loco/loco-regional recurrence is defined as cancer recurrence within the regional resection area or local anastomotic site.
  Distant recurrence is defined as peritoneal recurrence, liver metastasis or metastasis at other extra-abdominal sites as well as nodal metastasis beyond the regional nodes
Event-free survival (EFS) | up to 5 years; from the date of dostarlimab initiation to the date of surgery
  Event-free survival is defined as time from first dose of treatment to surgery for tumoral resection, first progression of disease local or distant recurrence, or death due to any cause. Alive patients without event will be censored at the last follow-up.
Time to treatment failure (TTF) | up to 5 years; from the date of dostarlimab initiation to the date of progression or death
  Time to treatment failure is defined as the interval between initiating therapy (first dose of dostarlimab) and the earliest of clinical progression, depending on whether the patient had surgery for tumoral resection or no, or death.
Disease-free survival (DFS) | up to 5 years; from the date of surgery to the date of recurrence or death from any cause
  Disease-free survival is defined only for patient with surgery (partial or complete gastrectomy or oesogastrectomy) as the time between the date of surgery and the date either of recurrence or death from any cause.
Overall survival (OS) | up to 5 years; from the date of dostarlimab initiation to the date of death
  Overall survival is defined as the time between the date of the first dose of study treatment and the death date.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Andre, MD, Principal Investigator — Saint-Antoine Hospital
Locations (2):
- France (2):
  - CHRU Lille, Lille
  - Hôpital Saint Antoine, Paris

IPD SHARING:
Plan to Share IPD: No